CLINICAL TRIAL: NCT04719169
Title: Comparison Study of MRI-Enema and Water Soluble Contrast Enema in the Assessment of Colorectal Anastomotic Integrity Prior to Stoma Reversal
Brief Title: MRI Anastomotic Integrity of Pelvic Intestinal Anastomoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: mrianastv1.327102016; 191029 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2018-04-16; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-02

CONDITIONS: Ulcerative Colitis; Ileal Pouch; Anastomotic Leak
MeSH Terms: conditions — Colitis, Ulcerative; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-low pelvic colorectal anastomosis (Experimental): Single armed study
  Interventions: Diagnostic Test: Dynamic MRI enema; Diagnostic Test: Fluoroscopic enema

INTERVENTIONS:
Diagnostic Test: Dynamic MRI enema — Dynamic MRI enema
Diagnostic Test: Fluoroscopic enema — Fluoroscopic enema

SUMMARY:
This protocol describes using an MRI-Enema technique to assess the integrity of colorectal anastomoses when compared to fluoroscopic water soluble contrast enema, and provides information the participant recruitment process, participant experience and study management.

DETAILED DESCRIPTION:
Both examinations will be performed ideally on the same day or a maximum of 7 days apart. The order of the two tests will be directed according to scan appointment availability. The WSCE will take place at St Marks Hospital London. Due to the MRI capacity at LNWH trust the MRI-Enema will take place at Number 9 Harley Street, London. A service level agreement will be in place for the scans to occur, and St Marks Seedcorn funding has already been awarded to fund the MRI scans. The patients will be asked to fill in a survey to assess their experience immediately after each test in each location.

MRI-Enema:

A 16Fr Foley catheter is introduced per-anus with the patient in a left lateral decubitus position on the MRI scanner table. If the anastomosis was low (within 5 cm of anorectal junction) the catheter will be taped to the skin to maintain its position. In the event of a mid-rectal or upper rectal anastomosis (>5 cm from anorectal junction), the catheter balloon may be filled with 2-5mls of water and withdrawn to a location at the top of the anal sphincter complex. In both instances, after catheter insertion the patient is then re-positioned to a supine body position.

The MRI protocol used is detailed below. In summary, T2 and T1 (with fat suppression) sequences are obtained prior to filling the lumen with contrast to assess the presence of any pre-sacral and peri-anastomotic fluid, to identify the presence of haematoma and to ensure the catheter is appropriately sited with the catheter tip above the anal canal and close to the anastomosis, ideally within 3cm.

The enema comprises a mixture of normal saline (400mls) and contrast agent (Gadovist, 4mls) to produce a 1% contrast solution which part fills a standard contrast enema bag and delivery system. The bag is attached to a fixed hook located 100cm above the scanner table height, such that fluid will deliver from the bag via the catheter according to gravity.

Dynamic MRI sequences are then performed with the delivery tube open to maximise flow of contrast into the residual rectum/neo-rectum or ileo-anal pouch.

Following the dynamic sequences, further axial and coronal images are acquired in order to identify the presence of leaked fluid within the pelvis.

After all images have been acquired, the enema bag is then placed on the floor to allow drainage of enema solution back into bag prior to removal of catheter.

MRI Protocol:

Pre Enema T2 sagittal Pre Enema T2 sagittal Fat-sat Pre Enema T2 axial SFOV Pre Enema T1 axial Filling Phase Dynamic sagittal Post Enema 3D volumetric T1 sagittal SFOV Post Enema T2 axial fat sat Post Enema T2 coronal fat sat

WSCE:

The WSCE is undertaken according to standard practice. As with the MRI, a 16Fr Foley catheter is introduced per anus with the patient in the left lateral decubitus position. Having affixed the catheter in place according to the height of the anastomosis above the anorectal junction as described above, water-soluble contrast (Gastrografin) is introduced via an enema delivery bag system as described above.

Radiographic images are then acquired with the patient in the supine and lateral decubitus positions as required in order to delineate the anastomosis and any related leak of contrast. The bag is then placed on the floor to allow drainage of fluid and the catheter removed.

Patients will be asked to complete a questionnaire immediately following both examinations. Questions will be targeted to evaluate anxiety, comfort, embarrassment and confidence in the test's outcome.

Reference standard = Consensus of both tests (WSCE and MRI-Enema) with agreement between two radiologists and in agreement with referring consultant /clinical assessment including findings at clinical examination where applicable.

ELIGIBILITY:
Inclusion Criteria:

1. History of colonic / anterior resection with low pelvic anastomosis including: ileorectal anastomosis, ileal pouch-anal anastomosis, colorectal anastomosis.
2. Clinical requirement for assessment of anastomotic integrity (e.g. prior to reversal of defunctioning stoma)
3. Ambulatory Patient
4. Over 18 years of age

Exclusion Criteria:

1. History of gadolinium allergy
2. Contraindication to MRI
3. Known inability to tolerate MRI (e.g. claustrophobia)
4. Known inability to maintain anal continence
5. Unable or unwilling to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
The test accuracy of (1) water-soluble contrast enema (WCSE) for the detection of colorectal anastomotic leaks. The reference standard will be consensus of Radiologist interpretation and surgical clinical assessment. | Up to 36 months
  As above
The test accuracy of (2) MRI-Enema for detection of colorectal anastomotic leaks. The reference standard will be consensus of Radiologist interpretation and surgical clinical assessment. | Up to 36 months
  As above

SECONDARY OUTCOMES:
(1) The comparative sensitivity for reported outcome variables relevant to investigation of pelvic intestinal anastomotic integrity. Including but not limited to: collection, fistula, fibrosis, lymphadenopathy, stenosis. | Up to 36 months
  As above
(2) Patient experience of WSCE vs MRI-Enema particularly relating to anxiety, comfort and embarrassment assessed on a non-validated five point questionnaire entitled 'MRI-Enema Study Patient Questionnaire v1.1'. | Up to 36 months
  13 statements are answered in tick boxes on a five-point scale categorised to: 'Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree'. For nearly all statements, agreement is a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- St Mark's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be available to members of the research team included in the study delegation log and members of the patient's normal clinical care team.

REFERENCES:
- [Derived] Worley G, Burling D, Corr A, Clark S, Baldwin-Cleland R, Faiz O, Jenkins J. MRI-enema for the assessment of pelvic intestinal anastomotic integrity. Colorectal Dis. 2021 Jul;23(7):1890-1899. doi: 10.1111/codi.15688. Epub 2021 May 16. PMID 33900000